CLINICAL TRIAL: NCT01760382
Title: REgister of Myocardial Infarction Patients Treated by the NOVAra STE-MI Network
Acronym: RENOVAMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, Principal investigator, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: RENOVAMI01
Record Dates: First submitted 2012-12-30; First posted 2013-01-04 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; ST elevation myocardial infarction; primary PCI; reperfusion therapy; angioplasty; stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- STEMI network Primary PCI patients: Patients with STEMI brought to the Hub Hospital by the STEMI network ambulance and treated by primary PCI.
  Interventions: Device: Primary PCI
- STEMI Hospital ED Primary PCI patients: Patients with STEMI who reached by themselves the Hub Hospital, where they were admitted for STEMI and tretated by Primary PCI
  Interventions: Device: Primary PCI

INTERVENTIONS:
Device: Primary PCI — mechanical reopening of the STEMI-related coronary artery by PTCA, with or without coronary stent implantation

SUMMARY:
Myocardial infarction (MI) outcomes strictly depend on the time to reponed the infarct-related coronary artery. Networks have been activated in the last years in many countries to achieve fast track access of patients with ST-elevation MI to hospital with h24 primary PCI availability or directly to Cath Labs. From 2011 a regional STEMI network have been formally activated in Piedmont. The aim of our registry is to monitor the activity of the STEMI network in the large suburban area of Novara (population of about 800.000 subjects).

DETAILED DESCRIPTION:
Myocardial infarction (MI) outcomes strictly depend on the time to reponed the infarct-related coronary artery. Networks have been activated in the last years in many countries to achieve fast track access of patients with ST-elevation MI to hospital with h24 primary PCI availability or directly to Cath Labs. From 2011 a regional STEMI network have been formally activated in Piedmont. The aim of our registry is to monitor the activity of the STEMI network in the large suburban area of Novara (population of about 800.000 subjects).

Novara STEMI network depends on the 118 service (the same of 911 in USA). When a call for suspected MI is processed, an Ambulance capable of transmitting a 12D ECG to the Hub Center is sent to the patient domicile. If the ECG and history suggest STEMI and transport time <90min, the patient is given aspirin and sent to Hub Hospital for primary PCI. If transport time is estimated >90min thrombolysis with TNK is performed in ambulance and the patient is sent to Hub Hospital for rescue PCI or re-evaluation in case of reperfusion.

Inclusion criteria: all patients with STEMI admitted to Novara Hospital (3rd level Hub with Cardiac Surgery Facility). No exclusion criteria.

Patients will be divided for comparisons in 2 groups (Group A: people admitted to hospital through the STEMI network. Group B: people admitted for STEMI through the Emergency department of the Novara Hospital or via secondary trasports regulated by Spoke Hospitals).

Quality factors: recording of time from symptoms onset and 1st medical contact, time from 1st medical contact and coronary angiography (door to needle time) and time from 1st medical contact and mechanical reperfusion (door to balloon time), angiographic indexes of reperfusion (baseline and postprocedural TIMI flow, blush grade, corrected TIMI frame count), trends for ST elevation resolution,trends for troponin and CK-MB dismission, baseline and postprocedural echocardiography. Clinical outcomes will be successful reperfusion, in-hospital cardiac mortality, in-hospital reinfarction and in-hospital stent thrombosis. Moreover patients will be followed up clinically for at least 1 year (outcomes: cardiac mortality, reinfarction, symptoms/ischemia driven target vessel revascularization).

ELIGIBILITY:
Inclusion Criteria:

* chest pain or equivalents (dyspnea, epigastrial pain) within 12 hours from onset (also after 12 hours if patient still symptomatic)
* ST segmnent elevation on more 2 or more contiguous ECG leads
* reperfusion treatment by primary PCI

Exclusion Criteria:

* symptoms beginning more than 12 hours before (with patient asymptomatic)
* survival estimated < 6 months according to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest pain or equivalents (dyspnea, epigastrial pain) and ST segmnent elevation on more 2 or more contiguous ECG leads
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Successful reperfusion | 1 day
  Successful reperfusion of the infarct related artery according to both clinical (>70% reduction of ST elevation 90min after primary PCI, in comparison to baseline) and angiographic criteria (restoration of TIMI 3 flow with blush grade at least 2).

SECONDARY OUTCOMES:
In Hospital Cardiac Mortality | 1 week
  In Hospital death for cardiac causes
In hospital myocardial infarction | 1 week
  In hospital new myocardial infarction described as new episode of chest pain with new q waves on ECG and/or new release (secondary peak) of troponin/CK-MB
In hospital stent thrombosis | 1 week
  In hospital thrombosis of the stent implanted in the STEMI-related artery

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, M.D., Principal Investigator — Azienda Ospedaliero Universitaria Maggiore della Carita
Locations (1):
- Azienda Ospedaliero Universitaria Maggiore della Carita, Novara, Piedmont, Italy

REFERENCES:
- [Derived] Lupi A, Bona RD, Meliga E, Capodanno D, Schaffer A, Bongo AS, Gaudio G, Guasti L, Alexopoulos D, Valgimigli M, Porto I. Early P2Y12 Inhibitors Escalation in Primary PCI Patients: Insights from the RENOVAMI Registry. Thromb Haemost. 2018 May;118(5):852-863. doi: 10.1055/s-0038-1635578. Epub 2018 Apr 4. PMID 29618159